CLINICAL TRIAL: NCT06787872
Title: PREVALENCE of LICHEN PLANUS AMONG PATIENTS REFERRED to the DEPARTMENT of ORAL DISEASES and PERIODONTOLOGY, LJUBLJANA, SLOVENIA in the PERIOD 2021-2023
Brief Title: Prevalence of Lichen Planus
Status: Completed | Type: Observational
Sponsor: University of Ljubljana (Other)
Responsible Party: Sponsor
Other Study IDs: Oral lichen planus prevalence
Record Dates: First submitted 2025-01-16; First posted 2025-01-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Oral Lichen Planus
MeSH Terms: conditions — Lichen Planus, Oral

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Clinical records of all patients referred to the Department of Oral diseases and periodontology in the period 2021-2023 were retrogradely assesed. The prevalence of patients with the diagnosis of Oral lichen planus and contributing factors were accordingly analyzed.

DETAILED DESCRIPTION:
Clinical records of 111 patients with the clinical or histopathological diagnosis of Oral ichen planus were included in the study. The prevalence of oral lichen planus was calculated and all the contributing factors including age, gender, location, type, skin involvement, presence of peridontal disease, systemic diseases and medications were assesed.

ELIGIBILITY:
Inclusion Criteria:

* All patients clinically or histopathologically diagnosed with Oral Lichen Planus

Exclusion Criteria:

* All patients not clinically or histopathologically diagnosed with Oral Lichen Planus

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 111 patients with Oral Lichen Planus referred to the Departement of Oral diseases and Periodontology, Ljubljana, Slovenia during the period 2021-2023 were included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Prevalence of Oral Lichen Planus of referred patients | 2021-2023
  Prevalence of Oral Lichen Planus of referred patients to the Departement of Oral diseases and periodontology in the period 2021-2023 was assesed.

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Centre, Ljubljana, Slovenia, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No
The IPD will not be shared due to privacy of the patients